CLINICAL TRIAL: NCT04779216
Title: Effects of Romosozumab on Bone Density, Markers of Bone Metabolism and Bone Microarchitecture in Women With Anorexia Nervosa: A Pilot Study
Brief Title: Effects of Romosozumab on Bone Density in Women With Anorexia Nervosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karen Klahr Miller, MD (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Karen Klahr Miller, MD, Professor of Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P000329
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Bone Density, Low; Bone Loss; Anorexia Nervosa; Eating Disorders
MeSH Terms: conditions — Bone Diseases, Metabolic; Anorexia Nervosa; Feeding and Eating Disorders | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Romosozumab 210mg Injection (Experimental): Romosozumab 210mg injection monthly for 12 months. A single infusion of open-label zoledronic acid 5 mg after the initial 12-month administration of romosozumab.
  Interventions: Drug: Romosozumab Prefilled Syringe; Drug: Zoledronic acid 5 mg
- Placebo (Placebo Comparator): Placebo injection monthly for 12 months. A single infusion of open-label zoledronic acid 5 mg after the initial 12-month administration of placebo.
  Interventions: Drug: Placebo; Drug: Zoledronic acid 5 mg

INTERVENTIONS:
Drug: Romosozumab Prefilled Syringe — Romosozumab 210mg Injection monthly for 12 months
  Arms: Active Romosozumab 210mg Injection
Drug: Placebo — Placebo Injection monthly for 12 months
  Arms: Placebo
Drug: Zoledronic acid 5 mg — A single infusion of open-label zoledronic acid 5 mg after the initial 12-month administration of romosozumab or placebo
  Other Names: Zoledronate, Reclast

SUMMARY:
This protocol is a randomized, double-blind, placebo-controlled clinical trial which aims to investigate the effect of romosozumab on BMD in women with anorexia nervosa. The investigators will also investigate the safety of romosozumab in women with anorexia nervosa. The investigators hypothesize that 12 months of romosozumab administration will result in an increase in bone mineral density, increase in markers of bone formation and decrease in markers of bone resorption, and improvement in bone microarchitecture in osteopenic women with anorexia nervosa compared with placebo.

In Phase 2, participants will receive a single infusion of open-label zoledronic acid (an intravenous bisphosphonate) 5 mg after the initial 12-month administration of romosozumab or placebo. The investigators hypothesize that 12 months of romosozumab followed by a single intravenous infusion of open-label zoledronic acid will result in a greater increase in BMD compared to 12 months of placebo followed by a single intravenous infusion of open-label zoledronic acid. Within the group of women who receive sequential therapy with 12 months of romosozumab followed by a single intravenous infusion of zoledronic acid, the investigators hypothesize BMD will be maintained between 12 and 24 months following administration of zoledronic acid.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 20-60 years, skeletally mature with closed epiphyses
* Body mass index (BMI) ≥ 16.5 kg/m2
* Anorexia nervosa or atypical anorexia nervosa defined by DSM-V diagnostic criteria
* BMD Z-score < -1.0
* Normal serum 25-OH vitamin D (>30 ng/mL) and calcium levels
* For women of reproductive age, agree to use an effective contraceptive method. Highly effective methods of birth control include: Combined (estrogen and progestogen) hormonal methods (pills, vaginal ring, or skin patch); Intrauterine device (IUD); Intrauterine hormonal-releasing system (IUS); Surgery to tie both fallopian tubes (bilateral tubal ligation/occlusion); Woman's male partner has had a vasectomy and testing shows there is no sperm in the semen
* Dental check-up within the past year

Exclusion Criteria:

* Hospitalization within 3 months of baseline study visit, including inpatient eating disorder treatment facility; participating in a residential eating disorder treatment program within 3 months of study participation is permitted
* Myocardial infarction or stroke within 1 year preceding enrollment
* History of hypertension or use of anti-hypertensive medications within the past 6 months
* Any disease known to affect bone, including untreated thyroid dysfunction, Cushing's or renal failure
* Any medication known to affect bone metabolism within 3 months of the study, excluding oral contraceptives or other forms of estrogen administration. Bisphosphonates must have been discontinued for at least one year before participation
* Immunodeficiency or taking immunosuppressive therapy
* Serum 25-OH vitamin D level <30 ng/mL
* Serum potassium <3.0 meq/L
* Serum magnesium <1.5 meq/L
* Serum ALT >3 times upper limit of normal
* eGFR of less than 30 ml/min
* LDL > 190 mg/dL
* Hypocalcemia
* Diabetes mellitus
* Active substance abuse, including alcohol
* Current smoker
* History of malignancy
* Paget disease of bone
* Osteomalacia
* Osteonecrosis of the jaw (ONJ) or risk factor for ONJ, such as invasive dental procedures (eg, tooth extraction, dental implants, oral surgery in the past 6 months), poor oral hygiene, periodontal and/or pre-existing dental disease, and current use of corticosteroids.
* Planned invasive dental procedure over the next 24 months
* Known sensitivity to any of the products or components of the medication to be administered
* Sensitivity to calcium or vitamin D supplements
* Pregnant, planning to become pregnant within 12 months after the end of treatment and/or breastfeeding
* Hypersensitivity to any component of zoledronic acid

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, double-blind, placebo-controlled trial. 30 subjects randomized in a 2:1 ratio to romosozumab followed by zoledronic acid or placebo followed by zoledronic acid
Groups:
- Active Romosozumab 210mg Injection: Romosozumab 210mg injection monthly for 12 months. A single infusion of open-label zoledronic acid 5 mg at the 12-month visit.
- Placebo: Placebo injection monthly for 12 months. A single infusion of open-label zoledronic acid 5 mg at the 12-month visit.
Period: Overall Study
Arm/Group | Active Romosozumab 210mg Injection | Placebo
Started | 20 | 10
Completed | 18 | 10
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Romosozumab 210mg Injection: Romosozumab 210mg Injection monthly for 12 months
  A single infusion of open-label zoledronic acid 5 mg at the 12-month visit.
- Total: Total of all reporting groups
Arm/Group | Active Romosozumab 210mg Injection | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (13) | 27 (6) | 31 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 9 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 8 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Postero-anterior (PA) lumbar spine bone mineral density (BMD) Mean (Standard Deviation) [Mean (Standard Deviation); unit: g/cm^2] | 0.84 (0.092) | 0.81 (0.065) | 0.83 (0.084)
Postero-anterior (PA) lumbar spine BMD Z-score [Mean (Standard Deviation); unit: Z-score] — PA lumbar spine BMD Z-score was obtained by dual-energy x-ray absorptiometry (DXA). A BMD Z-score is the number of standard deviations above or below the mean BMD given a person's age, sex, and race. A BMD Z-score of "0" represents the population mean. A BMD Z-score >0 represents a higher/better BMD, whereas a BMD Z-score <0 represents a lower/worse BMD.
  Z-score | -1.60 (0.88) | -2.06 (0.60) | -1.75 (0.82)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: One subject's BMI was adjusted for amputation.
  kg/m^2 | 19.3 (2.2) | 18.8 (1.2) | 19.1 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to 12 Months in Postero-anterior Lumbar Spine Bone Mineral Density by Dual Energy X-ray Absorptiometry (DXA).
Description: Percent change from baseline to 12 months in postero-anterior lumbar spine bone mineral density by dual energy x-ray absorptiometry (DXA).
Time Frame: Baseline to 12 Months
Population: Women, age 20-60 years, with anorexia nervosa
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Active Romosozumab 210mg Injection | Placebo
Number analyzed (Participants) | 20 | 10
% change | 12.4 (4.2) | -0.3 (3.7)
Statistical Analysis 1: Comparison: Active Romosozumab 210mg Injection vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Secondary Outcome: Percent Change From Baseline to 24 Months in Postero-anterior Lumbar Spine BMD.
Description: Percent change from baseline to 24 months in postero-anterior lumbar spine bone mineral density (BMD) by dual energy x-ray absorptiometry (DXA). This is a secondary endpoint at 24 months (study completion). The 24-month completion date was 11/17/2025. The 24-month results will be reported in November 2026.
Time Frame: Baseline to 24 Months
Reporting Status: Not Posted, anticipated posting 2026-11

ADVERSE EVENTS:
Time Frame: Baseline to 12 months.
Arm/Group | Active Romosozumab 210mg Injection | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 12/20 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Romosozumab 210mg Injection (N=20) | Placebo (N=10)
Irritation/soreness/swelling at injection sites (Skin and subcutaneous tissue disorders) | 8 | 1
COVID-19 (Infections and infestations) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Headache (General disorders) | 2 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Intermittent galactorrhea (Reproductive system and breast disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/16/NCT04779216/Prot_SAP_000.pdf